CLINICAL TRIAL: NCT00456144
Title: Prospective Observation Study of Insulin Sensitivity During and After Gonadotropin Releasing Hormone (GnRH) Agonist Therapy for Prostate Cancer
Brief Title: Prospective Observation Study of Insulin Sensitivity During and After Gonadotropin Releasing Hormone Agonist Therapy for Prostate Cancer
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Matthew R. Smith, MD, PhD, Director, Genitourinary Malignancies Program, Massachusetts General Hospital
Other Study IDs: 06-086
Record Dates: First submitted 2007-04-02; First posted 2007-04-04 (Estimated); Last update posted 2013-07-11 (Estimated); Status verified 2013-07

CONDITIONS: Prostate Cancer
Keywords: GnRH; Insulin sensitivity
MeSH Terms: conditions — Prostatic Neoplasms; Insulin Resistance

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood Urine

GROUPS / COHORTS (2):
- Group 1: GnRH agonist for 24 months
  Interventions: Drug: Gonadotropin Releasing Hormone Agonist Therapy
- Group 2: GnRH agonist for 6 months
  Interventions: Drug: Gonadotropin Releasing Hormone Agonist Therapy

INTERVENTIONS:
Drug: Gonadotropin Releasing Hormone Agonist Therapy — Given either for 24 months and 6 months

SUMMARY:
The purpose of this research study is to find out if a certain type of hormone therapy, gonadotropin-releasing hormone agonist (GnRH agonist), affects the way the body produces and responds to insulin. The investigators will evaluate the changes in insulin sensitivity during and after GnRH agonist treatment for prostate cancer. The investigators are assessing the possibility that treatment-related insulin resistance may contribute to the risk of diabetes and/or cardiovascular disease in men with prostate cancer.

DETAILED DESCRIPTION:
* The study will be divided into 2 groups: one group (Cohort A) will consist of men undergoing GnRH agonist therapy for at least 24 months. The second group (Cohort B) will consist of men undergoing the same treatment but who are scheduled to receive only 6 months of treatment.
* The following tests and procedures will be performed when the participant joins the study, then at 3, 6, 12 and 24 months thereafter. (All visits will take place at the General Clinical Research Center (GCRC) at the Massachusetts General Hospital.) Height and weight; blood and urine samples; Oral Glucose Tolerance Test (OGTT), Dual energy X-ray Absorptiometry scan; medical history; and physical examinations.

ELIGIBILITY:
Inclusion Criteria:

* Adenocarcinoma of the prostate, clinical stage M0
* Scheduled to initiate GnRH agonist therapy with intended treatment duration of greater than 24 months (Group A)
* Scheduled for radiation therapy and neoadjuvant GnRH agonist therapy with intended 6 month duration of treatment (Group B)
* Karnofsky Performance Status 90 or 100
* Local or local-regional disease (Group B)

Exclusion Criteria:

* Prior hormone therapy (GnRH agonist or antiandrogen)
* History of bilateral orchiectomy
* Known diabetes mellitus or glucose intolerance
* Current treatment with anabolic agents or metabolic agents known to affect insulin or glucose levels

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men with prostate cancer scheduled to undergo GnRH agonist therapy with intended treatment duration of 6 or 24 months.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2006-08; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew R. Smith, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Result] Saylor PJ, Karoly ED, Smith MR. Prospective study of changes in the metabolomic profiles of men during their first three months of androgen deprivation therapy for prostate cancer. Clin Cancer Res. 2012 Jul 1;18(13):3677-85. doi: 10.1158/1078-0432.CCR-11-3209. Epub 2012 May 15. PMID 22589396